CLINICAL TRIAL: NCT01176760
Title: The Significances of Intact Vagal Innervation for the Glucose and GLP1 Induced Insulin Secretion
Brief Title: Intact Vagal Innervation for and Glucagon-like Peptide-1 (GLP-1) Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jonatan I Bagger, MD, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Truncated isoglycemia
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Vagotomy, Truncal
Keywords: vagotomy; vagus; GLP-1; Insulin secretion
MeSH Terms: interventions — Dipeptidyl Peptidase 4; Vildagliptin; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vago (Experimental): Truncally vagotomized subjects (due to duodenal ulcer operation)
  Interventions: Drug: Dipeptidyl peptidase 4 (DPP 4) inhibitor; Other: oral glucose
- Cardia (Experimental): Truncally vagotomized subjects (due to cardia resection)
  Interventions: Drug: Dipeptidyl peptidase 4 (DPP 4) inhibitor; Other: oral glucose
- Ctrl (Experimental): Healthy matched control subjects
  Interventions: Drug: Dipeptidyl peptidase 4 (DPP 4) inhibitor; Other: oral glucose

INTERVENTIONS:
Drug: Dipeptidyl peptidase 4 (DPP 4) inhibitor — One tablet (50 mg)of DPP4 inhibitor is to be taken 12 and 1 hours before start of the oral glucose tolerance test (50 g glucose and 1.5 g paracetamol dissolved in 300 ml water)on day 3
  Other Names: Galvus
Other: oral glucose — 50 g glucose dissolved in 300 ml water with 1,5 g paracetamol is to be ingested orally within the first 15 minutes.
  Other Names: panodil

SUMMARY:
The aim of this study is to investigate the role of transmission via the vagal nerve for the effect of glucose and Glucagon-like peptide-1 (GLP-1) in respect to insulin secretion.

The hypothesis is that a great deal of the effects of GLP-1 is mediated via the nervous system and for this reason the investigators will research individuals with and without intact nervous supply.

DETAILED DESCRIPTION:
GLP-1 is a potent enterogastron and incretin hormone. It is rapidly inactivated by dipeptidyl peptidase IV so only 10-15% enters the systemic circulation. This has led to the hypothesis that GLP-1 interact locally with afferent sensory nerve fibers. We investigated the role of intact vagal innervations on the effect of glucose and GLP-1 on the insulin secretion

ELIGIBILITY:
Inclusion Criteria:

* normal fasting plasma glucose
* normal hemoglobin
* informed consent

Exclusion Criteria:

* type 1 diabetes mellitus or type 2 diabetes mellitus
* body mass index > 30
* inflammatory bowel disease
* intestinal surgery
* serum creatinine > 250 µM and/or albuminuria
* ALAT > 2 x normal value
* Severe cardiac insufficiency
* in treatment with medicine which cannot be paused for 12 hours

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
insulin secretion | four hours
  The insulin secretion during a four-hour oral glucose tolerance test (OGTT) and an intravenous isoglycaemic clamp is evaluated

SECONDARY OUTCOMES:
plasma GLP-1 | 12 time points within four hours
  12 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour
plasma GIP | 12 time points within four hours
  12 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour
plasma glucagon | 12 time points within four hours
  12 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour
plasma GLP-2 | 12 time points within four hours
  12 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour
plasma PYY | 12 time points within four hours
  12 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Plamboeck, MD, Principal Investigator — University Hospital, Gentofte, Copenhagen; Tina Vilsbøll, MD, dr.med, Study Director — University Hospital, Gentofte, Copenhagen
Locations (1):
- Department of internal medicine F´laboratory, Gentofte Hospital, Hellerup, Copenhagen, Denmark

REFERENCES:
- [Derived] Plamboeck A, Veedfald S, Deacon CF, Hartmann B, Wettergren A, Svendsen LB, Meisner S, Hovendal C, Knop FK, Vilsboll T, Holst JJ. Characterisation of oral and i.v. glucose handling in truncally vagotomised subjects with pyloroplasty. Eur J Endocrinol. 2013 Jul 6;169(2):187-201. doi: 10.1530/EJE-13-0264. Print 2013 Aug. PMID 23704713